CLINICAL TRIAL: NCT05374980
Title: The Effects of Fermented Milk Product With Probiotic on Helicobacter Pylori Infection, Gut Microbiome and Metabolism.
Brief Title: The Effects of Yogurt on Gut Microbiome and Metabolism in H. Pylori.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Han-Chung, Lien, Principle Investigator of Gastrointestinal Motility Lab, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SF19354B
Record Dates: First submitted 2022-04-13; First posted 2022-05-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Probiotic; Gut Microbiota; Helicobacter Pylori Infection; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yogurt (Experimental): Drink a bottle of 200ml yogurt every morning and evening for 8 weeks
  Interventions: Dietary Supplement: Yogurt
- Placebo (Placebo Comparator): Drink a bottle of 200ml placebo every morning and evening for 8 weeks
  Interventions: Dietary Supplement: Placebo
- Healthy volunteer (No Intervention): Patients with Helicobacter pylori negative (ΔUBT<2%) need blood test and collect stool samples at first, and collect stool samples again after 2 months.

INTERVENTIONS:
Dietary Supplement: Yogurt — Drink a bottle of 200ml yogurt every morning and evening for 8 weeks
  Arms: Yogurt
Dietary Supplement: Placebo — Drink a bottle of 200ml placebo every morning and evening for 8 weeks
  Arms: Placebo

SUMMARY:
Helicobacter pylori is a common pathogen causing upper gastrointestinal diseases including gastric ulcer and gastric cancer. Recent epidemiological findings have also shown that it is also related to colon cancer, metabolic syndrome, gut dysbiosis, glycemic control and insulin resistance.

The aim of this study is to investigate whether the gut microbiota and insulin resistance of patients with H. pylori infection are abnormal. In addition, whether drinking fermented milk product with probiotic reduces Helicobacter pylori, improves gut microbiota, and increases butyrate-producing bacteria and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 70 years old with positive Helicobacter pylori gastric C13 urea breath test (ΔUBT>10%).
2. Negative gastric Helicobacter (ΔUBT<2%) matching age, gender, and body mass index.

Exclusion Criteria:

1. Unhealthy habits or poor health status, including habitual smoking, alcoholism, polypharmacy or drug abuses.
2. Patients with acute diseases, such as respiratory tract infection, acute gastroenteritis.
3. In the past three months, those who have had dyspepsia but have not undergone gastroscopy, or have a history of active gastrointestinal ulcers and gastrointestinal bleeding.
4. Those who have had gastrointestinal cancer or have undergone gastrointestinal surgery.
5. Those who are unwilling to delay receiving Anti-H. pylori therapy.
6. Newly diagnosed cancer (except basal cell carcinoma) or cancer treatment in the past 5 years.
7. People who have had cardiovascular disease, respiratory disease, autoimmune disease, mental disease or other chronic diseases that are not well controlled, such as myocardial infarction or stroke, chronic obstructive pulmonary disease, inflammatory bowel disease, Schizophrenia.
8. Diabetes and those who are or need to take drugs.
9. Those who have used the following drugs in the past month: antibiotics, NSAIDs, obesity drugs, steroid therapy, proton pump inhibitors, bismuth agents.
10. In the past month, regularly consume the following foods (at least 2 times a week): probiotics, prebiotics, or any foods containing probiotics, dairy products (yogurt, cheese), Chinese medicine, kimchi, miso, honey, cranberry, spicy food.
11. Fecal occult blood positive, unexplained iron-deficiency anemia, weight increase or decrease by more than 5% within six months.
12. Abnormal liver function index (AST, ALT or ALP greater than 2 times the upper limit of normal), abnormal renal function index (eGFR less than 45 ml/min).
13. Pregnant or breast-feeding women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Change of gut Microbiome | Baseline to day 28 and day 56
  uses high-throughput sequencing to sequence the 16S rRNA

SECONDARY OUTCOMES:
Change of C13 urea breath test | Baseline to day 28 and day 56
  Delta urea breath test

OTHER OUTCOMES:
Change of weight | Baseline to day 28 and day 56
  weight in kilograms
Change of waist circumference | Baseline to day 28 and day 56
  waist in centimeters
Change of blood pressure | Baseline to day 28 and day 56
  Change of systolic blood pressure and diastolic blood pressure
Change of HOMA-IR | Baseline to day 28 and day 56
  Glucose and insulin will be combined to report HOMA-IR in (mg/dl x mIU/L)/405
Change of high density lipoprotein | Baseline to day 28 and day 56
  Change of high density lipoprotein in the blood
Change of low density lipoprotein | Baseline to day 28 and day 56
  Change of low density lipoprotein in the blood
Change of Cholesterol | Baseline to day 28 and day 56
  Change of Cholesterol in the blood
Change of Triglyceride | Baseline to day 28 and day 56
  Change of Triglyceride in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Han-Chung Lien, MDPHD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cover TL, Blaser MJ. Helicobacter pylori in health and disease. Gastroenterology. 2009 May;136(6):1863-73. doi: 10.1053/j.gastro.2009.01.073. Epub 2009 May 7. PMID 19457415
- [Result] Sugizaki K, Tari A, Kitadai Y, Oda I, Nakamura S, Yoshino T, Sugiyama T. Anti-Helicobacter pylori therapy in localized gastric mucosa-associated lymphoid tissue lymphoma: A prospective, nationwide, multicenter study in Japan. Helicobacter. 2018 Apr;23(2):e12474. doi: 10.1111/hel.12474. Epub 2018 Mar 4. PMID 29504247
- [Result] Butt J, Varga MG, Blot WJ, Teras L, Visvanathan K, Le Marchand L, Haiman C, Chen Y, Bao Y, Sesso HD, Wassertheil-Smoller S, Ho GYF, Tinker LE, Peek RM, Potter JD, Cover TL, Hendrix LH, Huang LC, Hyslop T, Um C, Grodstein F, Song M, Zeleniuch-Jacquotte A, Berndt S, Hildesheim A, Waterboer T, Pawlita M, Epplein M. Serologic Response to Helicobacter pylori Proteins Associated With Risk of Colorectal Cancer Among Diverse Populations in the United States. Gastroenterology. 2019 Jan;156(1):175-186.e2. doi: 10.1053/j.gastro.2018.09.054. Epub 2018 Oct 6. PMID 30296434
- [Result] Park H, Park JJ, Park YM, Baik SJ, Lee HJ, Jung DH, Kim JH, Youn YH, Park H. The association between Helicobacter pylori infection and the risk of advanced colorectal neoplasia may differ according to age and cigarette smoking. Helicobacter. 2018 Jun;23(3):e12477. doi: 10.1111/hel.12477. Epub 2018 Mar 29. PMID 29600573
- [Result] Chen TP, Hung HF, Chen MK, Lai HH, Hsu WF, Huang KC, Yang KC. Helicobacter Pylori Infection is Positively Associated with Metabolic Syndrome in Taiwanese Adults: a Cross-Sectional Study. Helicobacter. 2015 Jun;20(3):184-91. doi: 10.1111/hel.12190. Epub 2015 Jan 12. PMID 25582223